CLINICAL TRIAL: NCT04179370
Title: The Relationship Between Sun Exposure, Diet, Lifestyle and Bone on Vitamin D Status (25OHD) in British African-Caribbean Women Living in Southern United Kingdom
Brief Title: Vitamin D and Health Status of British African-Caribbean Women
Status: Recruiting | Type: Observational
Sponsor: University of Surrey (Other)
Responsible Party: Sponsor
Other Study IDs: SPON 2019 025 FHMS
Record Dates: First submitted 2019-11-20; First posted 2019-11-27 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Vitamin D Deficiency
Keywords: vitamin D OR 25(OH)D; African-Caribbean OR Afro-Caribbean
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — A blood sample will be taken from participants and will include:
  * serum 25OHD, calcium and albumin, P1NP, CTX, lipid profile, micronutrient status
  * PTH plasma, blood glucose level
  * Whole Blood DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: N/A - no intervention. Observational study. — N/A - no intervention. Observational study.

SUMMARY:
Vitamin D deficiency remains a global public health issue (Wilson 2017). In the United Kingdom (UK). There is a lack of research looking at vitamin D status of the British African-Caribbean population. This population is particularly at risk to vitamin D deficiency due to possessing a skin type which hinders the production of vitamin D in the skin. Further, due to the geographical location of the UK, there is reduced ability to produce vitamin D due to the low sun exposure (Libon 2013 ). Our main source of vitamin D is through skin exposure to the sun. In the UK, the UV radiation is only strong enough in April-September (Wilson 2017) for the production of vitamin D to occur. In winter months, vitamin D needs to be consumed in food or supplement form. Vitamin D is essential for healthy bones and is associated with reduced risk of certain cancers and immune disorders (Wilson 2017). There is strong epidemiological evidence linking low vitamin D status with diabetes, cardiovascular disease, osteoporosis, osteoarthritis and some cancers (NatCen 2018).

This observational study will aim to determine the vitamin D status of British Afro-Caribbean women, as well as determine the effects of sun exposure, dietary vitamin D intake, muscular strength, lifestyle and anthropometrical (height, weight etc.) factors have on vitamin D status. The study will be conducted at the University of Surrey. The study will take place in Autumn and winter 2019/2020 and a repeat study in Spring 2020. Each participant will require two visits to the university, each session will take approximately 2 hours. The study is funded by the University of Surrey. The findings of this study may lead to strategies for improving vitamin D status in this population, as well as improving guidelines to assist darker-skinned people regarding sunlight exposure in high latitudes.

DETAILED DESCRIPTION:
Introduction

Vitamin D deficiency remains a global public health issue (Wilson 2017). There is strong epidemiological evidence linking low vitamin D status with diabetes, cardiovascular disease, osteoporosis, osteoarthritis and some cancers (NatCen 2018). The condition has a significant financial impact on the economy, therefore is of public health importance (Sturges 2018).

The British African-Caribbean population in the United Kingdom (UK) is steadily increasing (2011 UK census). Despite this, there is a lack of research looking at the vitamin D status of this population. This population is particularly at risk to vitamin D deficiency due to possessing a skin type which hinders the production of vitamin D in the skin (Libon 2013). Further, due to the geographical location of the UK, there is an even greater reduced ability to produce vitamin D due to the low sun exposure (Libon 2013).

Our main source of vitamin D is through skin exposure to the sun. In the UK, the UV radiation is only strong enough between April and September, for the production of vitamin D to occur (Wilson 2017). In winter months, vitamin D needs to be consumed in food or supplement form. Our study will look at the vitamin D status of British African-Caribbean women living in the UK in late autumn and winter 2019/2020 and compare these findings to a second sample in spring 2020. In addition, the investigators will determine which factors such as dietary intake, sun exposure and muscular strength contribute to vitamin D status. Each participant will require two visits to the university, the first session will take approximately 2 hours, while the second session will be shorter as not all measures will be repeated. The study is funded by the University of Surrey.

The findings of this study may lead to strategies for improving vitamin D status in this population, as well as improving guidelines to assist darker-skinned people regarding sunlight exposure in high latitudes.

Aims

Primary objectives:

1. Assess vitamin D status in British African-Caribbean women 18-35 and >55 years old
2. To compare vitamin D status of participants in late autumn and winter 2019/2020 to levels in spring 2020
3. Determine the effects of sun exposure, dietary vitamin D intake, muscular strength, lifestyle and anthropometric factors have on vitamin D status

   Secondary objectives:
4. Assess level of vitamin D consumption from diet
5. Measure bone mineral density, bone mineral composition and body composition
6. Assess level of physical activity
7. Measure level of UVB sun exposure
8. Measure muscular strength and endurance
9. Assess qualitatively the attitudes and behaviours around sun exposure
10. Compare data to previously collected data on Caucasian and South Asian populations

Hypothesis:

It is hypothesised that British African-Caribbean women will have poorer vitamin D status than their Caucasian counterparts. It is assumed that those with higher sun exposure and vitamin D dietary intake will have higher levels of vitamin D as well as stronger bone mineral density and muscular strength.

Criteria for participant selection:

Inclusion

* Women
* British African-Caribbean

  * Self-reported
  * Having African ancestral origin and migrated via the Caribbean islands, or having at least one parent with African ancestral origin that migrated via the Caribbean
* Living in England for >2 months
* Aged 18-35 or >55 years
* No significant health issues
* Pre-menopausal (regular menstrual periods) or Post-menopausal (menstrual periods stopped for longer than 12 consecutive months)
* BMI 18-30kg/m2

Exclusion

* Women in perimenopause or menopause
* Pregnant or planning pregnancy during study period
* Hypercalcaemia (>2.5mmol/L) - assessed and excluded at baseline
* Currently receiving treatment for medical conditions that are likely to affect vitamin D metabolism (osteoporosis, hormone replacement therapy, anti-estrogens treatment, antiepileptic drugs and breast cancer treatment)
* Regular use of sun beds
* Having a sun holiday one month prior to commencing study or plans for a sun holiday for more than 4 weeks within the study period
* Women who take vitamin D or calcium supplements (or multivitamin supplements that contain these vitamins) - If potential participant agrees to stop supplement use to join the study, a wash-out period of 8 weeks prior to commencing the study is acceptable
* Living in England for less than 2 months

Withdrawal

All participants will be notified during the consenting process that they are free to withdraw from the trial at any time, without giving a reason.

Number of participants to be recruited

The investigators will aim to recruit n = 100 participants to be included in the study in late autumn and winter 2019/2020, with these same participants coming to the repeat study in spring 2020.

This number is based on the minimum required to give reliable and generalisable results and be within financial and time constraints of the study.

Summary of experimental design and methods used

This is an observational study which will require two visits to the clinical investigation unit (CIU), at the University of Surrey, Guildford. One visit will take place in late autumn and winter 2019/2020 and the other in spring 2020.

Participants will be recruited through the National Health Services (NHS), local groups, community groups, university clubs and societies, flyers and social media. Those interested in the study will contact the researchers, and then will be sent a participant information sheet and a screening questionnaire to see if they meet inclusion criteria.

Recruited participants will come to CIU fasted. After signing a consent form the following measurements will be taken:

1. Anthropometric measurements The following anthropometrical measurements will be taken from each participant: Weight, height, waist to hip ratio, waist circumference, waist to height ratio and body composition.

   Weight and body composition will be measured to the nearest 0.1kg. This will be achieved using a Tanita Body Composition Analyser MC-180MA. Standing height will be measured using a wall stadiometer, to the nearest 0.1cm. Waist and hip circumference will be measured using a non-extendable standard measure tape, at the narrowest point of the torso for waist measurement (if this cannot be estimated, the level of the belly button will be used as a reference point), and the widest part of the hips for the hip measurement, to the nearest 0.1cm.

   Waist to hip ratio will be calculated by dividing the waist measurement by the hip measurement (waist ÷ hip) and the waist to height ratio will be calculated by dividing the waist measurement by the height measurement (waist ÷ height)
2. Blood sample An 8 hour-fasted blood sample will be taken by a trained phlebotomist.

   The following collection tubes will be used:
   * 15ml BD Vacutainer® SSTTM (red top) tube: serum 25OHD, calcium and albumin, P1NP, CTX, lipid profile, micronutrient status
   * 6ml BD Vacutainer® EDTA (purple) tube: PTH plasma, blood glucose level
   * 3ml EDTA: Blood DNA

   Blood sampling will occur once, at each of the two sessions. Approximately 25ml of blood will be taken during each of the sessions, with a total of 50ml of blood taken during the entire study.

   Albumin, lipid profile, micronutrient status and blood glucose level will be analysed at the University of Surrey. Bone markers; P1NP and CTX will be analysed at the Metabolic Bone Centre, Northern General Hospital, Sheffield. Serum 25OHD, PTH plasma, calcium will be analysed at the Imperial College healthcare NHS trust.

   Both the serum and plasma blood samples will be stored at -80°C at the University of Surrey.

   Following the blood sample participants will be provided with refreshments.
3. Peripheral computed tomography (pQCT) scan A pQCT scan will be taken to measure bone mineral composition. A scan of the non-dominant forearm will be performed. If the participant moves during the scan it will need to be repeated. The scan is painless and involves a very low total effective radiation dose of approximately 0.5 uSv.
4. Dual energy X-ray absorptiometry (DEXA) scan Prior to the DEXA scan, participants will take a pre-scan questionnaire, which includes declaring they are not pregnant. Participants will be given the option to take a pregnancy test before both the pQCT and DEXA scans.

   Two DEXA scans will be taken. One scan to assess whole body bone mineral density and body composition, and the other to specifically assess fracture risk by scanning the femoral the hip and femoral head. Effective exposure doses for these scans are approximately 9 uSv and 8 uSv respectively. Total research protocol dose is approximately 18 uSv, this is equivalent to approximately 3 days of natural background radiation.
5. Sit-to-stand test The 30 second Sit to Stand Test is used to measure leg strength and endurance. A chair without arms will be placed against a wall to prevent slipping. The participant will sit in the chair with their back straight, feet shoulder width apart on floor, with their arms crossed at their wrists and held against the chest. If the participant uses their arms to stand up they are scored 0. The participant will complete as many full stands as possible within 30 seconds.
6. Grip strength test The purpose of this test is to measure the maximum isometric strength of the hand and forearm muscles. Placing their arm at a right angle with the elbow at the side of the body, the participant will use their non-dominant hand to hold the hand grip dynamometer (5401 Hand Grip Dynamometer, Takei Scientific Instruments Co. Ltd, Niigata, Japan). The participant will squeeze the dynamometer with maximum effort for 5 seconds. An average of three tests will be taken, to the nearest 0.1kg.
7. International Physical Activity Questionnaire (IPAQ) short form A physical activity questionnaire will be undertaken to obtain data on physical activity in everyday lives.
8. Sun exposure questionnaire The sun exposure questionnaire measures how often participants spend in the sun across different seasons, what body parts were exposed and if they have been on a recent summer holiday.
9. Lifestyle questionnaire The lifestyle questionnaire measures a range of factors including skin type, medical history, education, behaviours and attitudes towards sun exposure and knowledge and consumption of vitamin D.
10. Instruction on how to complete a 4-day food diary 4-day food diaries will be kept to measure dietary intake, in particular, intake of vitamin D. These will be used at home for four days, one of which days will be a weekend day. The participants are asked to record the time, what they eat, method of cooking and the amount eaten. They will be instructed to send these back to the investigators using the freepost envelopes provided. The researchers may phone or email the participants if any further information of their diet is required. Data will be analysed using Nutritics® nutritional analysis software.
11. Instructions on how to wear a dosimeter to measure UVB exposure Participants will be asked to wear a dosimeter polysulphone film badge to measure UVB exposure. The dosimeters are clipped to the outer clothing with a pin, worn on the upper chest/shoulder region. Individuals are asked to wear the badge on from sunrise to sunset, for 4 days, one of which will be a weekend day. They are instructed to store the dosimeter in the supplied envelope (of thick and dark material to prevent further UVB exposure during storage) until returning.

Data will be read at the University of Surrey, prior and after dosimeter use. A Cecil Aquarius CE7200 Double Beam Spectophotometer (CV <1%) will be used at 330nm to detect a change in absorbency.

Results of individual badge doses are reported in standard erythema dose (SED) units (1 SED = 100 J/m2). To convert to SED the following formula will be used:

SED = 10.7 [∆a330] + 14.3 [∆a330]2 - 26.4 [∆a330]3 + 89.1 [∆a330]4 [∆a330] = Change in absorbance at 330nm of the dosimeter from pre- to post-UVB exposure

The participants will then be invited back to the CIU in spring 2020. At the second session, only the following measures will be repeated: Anthropometric measurements, blood sample, sit-to-stand test, grip-strength test, 4-day food diary and measurement of UVB exposure through wearing a dosimeter. The DEXA scan, pQCT scan and questionnaires will only be performed at the baseline session. The results from both visits will then be analysed.

Statistical Analysis Statistical analysis will be undertaken with support from the University of Surrey statistical department. All statistical analysis will be carried out using SPSS statistical software (version 25; SPSS Inc., Chicago, IL). Data will be checked for normality using appropriate testing. Appropriate parametric/non-parametric analysis will be applied.

Data Handling

Data will be handled by the principal investigator who will act as the custodian. The following guidelines will be followed:

* All data will remain confidential
* All participants will be given a unique study number, their personal information will never be referenced to
* Data will be coded with unique study number
* All anonymised data will be stored in a secure location on the University's servers and on password-protected computers
* Project data will be held for at least 6 years and all research data for at least 10 years in accordance with University policy and in accordance with the {UK} Data Protection Act (2018).
* When a subject does not meet the inclusion criteria, all questionnaires and collected data will be destroyed.

Study evaluation

Benefits to participants All participants in the study will be offered a summary of their results, including their vitamin D status and their bone density. DEXA scans are considered the gold standard method of measuring body composition, therefore valuable to participants. The participants will also gain important information on their vitamin D status, which they would not be able to receive unless they visited a GP for a blood test. Not only will these results be of interest to the participants, but the investigators will also ensure that the participants understand that they are contributing to the research in vitamin D in their population group, and their results may help to change guidelines, benefit future populations and produce effective public health campaigns. The participants will not be paid, however will be reimbursed for all travel expenses.

Risk to participants Subjects will require two visits to the University of Surrey, which may cause minor inconveniences, however subjects will be reimbursed for travel expenses.

The venepuncture may cause some minor discomfort, although the sample will be taken by an experienced phlebotomist to minimise any adverse effects. The peripheral Computed Tomography (pQCT) measurements (for assessment of bone mineral density) of the forearm are painless and involve a very low total radiation dose. If the participant moves during the scan it will need to be repeated. The doses received are very low, at approximately 0.5uSv. Therefore, the risks/adverse effects of the pQCT radiation are minimal. A total of two Dual energy X-ray absorptiometry (DEXA) scans, one for the assessment of whole-body bone mineral density and body composition, and the other to assess fracture risk by scanning the hip and femoral head will be performed. Effective exposure doses for these scans are approximately 9 uSv and 8 uSv respectively. The total research protocol dose is approximately 18 uSv. This is equivalent to approximately 3 days of natural background radiation. Based on this dose, this equates to total lifetime cancer risks of approximately 1 in 700,000 for participants aged 18-35 years (based on an average of 7.5% per Sv), and approximately 1 in 4,000,000 for participants aged >55 years (based on 1.5% per Sv) (Wall 2011).

The questionnaires (IPAQ, sunlight exposure and lifestyle) are unlikely to cause much inconvenience to women as they are brief and focused. The food diaries can be monotonous, but only last 4 days. The food diaries should not be of too much inconvenience as the women are asked to not change their usual eating habits and continue eating as they normally would. The dosimeters are non-invasive and are worn like a badge on the outside of clothing, this has been limited to 4 days. The sit-to-stand and grip-strength tests are simple tests that are unlikely to cause any fatigue or discomfort. Anthropometric measurements are unlikely to cause any stress or discomfort as they will be brief and non-invasive.

Benefits to scientific knowledge and public health policy

The longitudinal observation study will allow the analysis of change in vitamin D status of British African-Caribbean women. This will be of huge benefit as there is little known about the vitamin D status of this population. The findings of this study will not only fill this gap in the knowledge, but may also inform public health policy on vitamin D. The study will aim to determine which factors such as dietary vitamin D intake, sun exposure and muscular strength impact on vitamin D status in this population, which is little known. The study will also assess attitudes towards sun exposure, which may give insights that would be useful to inform public policy.

ELIGIBILITY:
Inclusion Criteria:

* Women
* British African-Caribbean Self-reported Having African ancestral origin and migrated via the Caribbean islands, or having at least one parent with African ancestral origin that migrated via the Caribbean
* Living in England for >2 months
* Aged 18-35 or >55 years
* No significant health issues
* Pre-menopausal (regular menstrual periods) or Post-menopausal (menstrual periods stopped for longer than 12 consecutive months)
* BMI 18-30kg/m2

Exclusion Criteria:

* Women in perimenopause or menopause
* Pregnant or planning pregnancy during study period
* Hypercalcaemia (>2.5mmol/L) - assessed and excluded at baseline
* Currently receiving treatment for medical conditions that are likely to affect vitamin D metabolism (osteoporosis, hormone replacement therapy, anti-estrogens treatment, antiepileptic drugs and breast cancer treatment)
* Regular use of sun beds
* Having a sun holiday one month prior to commencing study or plans for a sun holiday for more than 4 weeks within the study period
* Women who take vitamin D or calcium supplements (or multivitamin supplements that contain these vitamins) - If potential participant agrees to stop supplement use to join the study, a wash-out period of 8 weeks prior to commencing the study is acceptable
* Living in England for less than 2 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility based on gender
Study Population: The study population is women aged over 18, who are not in menopause. Healthy women who have African-Caribbean ancestry, and have lived in the UK for more than 2 months are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-02-07 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Vitamin D (serum 250HD) status | One measurement at baseline
  A blood sample will be taken from participants. This will be analysed using liquid chromatography tandem mass spectroscopy (LC-MS)
Change in vitamin D status | The first measurement will be performed in winter 2020, with a repeat measurement approximately 3 months later in spring 2020.
  A blood sample will be taken from participants. This will be analysed using liquid chromatography tandem mass spectroscopy (LC-MS)
Bone mineral composition | One measurement at baseline
  Peripheral computed tomography (pQct) scan
Dual energy X-ray absorptiometry (DEXA) of whole body | One measurement at baseline
  Assess bone mineral density
Dual energy X-ray absorptiometry (DEXA) of femoral head | One measurement at baseline
  Assess fracture risk
Change in blood bone marker | The first measurement will be performed in winter 2020, with a repeat measurement approximately 3 months later in spring 2020.
  P1NP (bone markers) will be measured from blood
Change in blood bone marker | The first measurement will be performed in winter 2020, with a repeat measurement approximately 3 months later in spring 2020.
  CTX (bone marker) will be measured from blood
Vitamin D intake | One measurement at baseline
  Vitamin D intake will be measured through a 4-day food diary which participants will fill out for 4 day at home after the study
Change in vitamin D intake | The first measurement will be performed in winter 2020, with a repeat measurement approximately 3 months later in spring 2020.
  Vitamin D intake will be measured through a 4-day food diary which participants will fill out for 4 day at home after the study
Sun exposure | One measurement at baseline
  sun exposure will be measured by a dosimeter which measures UVB exposure. Participants wear this like a badge, for 4 days after the study
Change in sun exposure from winter to spring | The first measurement will be performed in winter 2020, with a repeat measurement approximately 3 months later in spring 2020.
  sun exposure will be measured by a dosimeter which measures UVB exposure. Participants wear this like a badge, for 4 days after the study

SECONDARY OUTCOMES:
Anthropometrical measurements - weight | One measurement at baseline
  Weight (kg)
Anthropometrical measurements - change in weight | The first measurement will be performed in winter 2020, with a repeat measurement approximately 3 months later in spring 2020.
  measurement of weight (kg)
Anthropometrical measurements - height | One measurement at baseline
  measurement of standing height (cm)
Anthropometrical measurements - Hip circumference | One measurement at baseline
  measurement of hip (cm)
Anthropometrical measurements - waist circumference | One measurement at baseline
  measurement of waist (cm)
Anthropometrical measurements - change in waist circumference | The first measurement will be performed in winter 2020, with a repeat measurement approximately 3 months later in spring 2020.
  measurement of waist circumference (cm)
Anthropometrical measurements - change in hip circumference | The first measurement will be performed in winter 2020, with a repeat measurement approximately 3 months later in spring 2020.
  measurement of hip circumference (cm)
Blood analytes - calcium | One measurement at baseline
  Calcium (mg/dL)
Blood analytes - change in calcium levels | The first measurement will be performed in winter 2020, with a repeat measurement approximately 3 months later in spring 2020.
  Calcium (mg/dL)
Blood analytes - albumin | One measurement at baseline
  Albumin (g/dL)
Blood analytes - change in albumin levels | The first measurement will be performed in winter 2020, with a repeat measurement approximately 3 months later in spring 2020.
  Albumin (g/dL)
Blood analytes - lipid profile | One measurement at baseline
  lipid profile (mg/dL)
Blood analytes - change in lipid profile status | The first measurement will be performed in winter 2020, with a repeat measurement approximately 3 months later in spring 2020.
  lipid profile (mg/dL)
Blood analytes - PTH | One measurement at baseline
  Parathyroid hormone (PTH) (pg/mL)
Blood analytes - change in PTH levels | The first measurement will be performed in winter 2020, with a repeat measurement approximately 3 months later in spring 2020.
  Parathyroid hormone (PTH) (pg/mL)
Blood analytes - micronutrient status | One measurement at baseline
  micro nutrient status
Blood analytes - change in micronutrient status | The first measurement will be performed in winter 2020, with a repeat measurement approximately 3 months later in spring 2020.
  micro nutrient status
Blood analytes - blood glucose levels | One measurement at baseline
  Blood glucose level (mg/dL)
Blood analytes - change in blood glucose levels | The first measurement will be performed in winter 2020, with a repeat measurement approximately 3 months later in spring 2020.
  Blood glucose level (mg/dL)
Muscular strength - sit-to-stand test | One measurement at baseline
  sit-to-stand test (number of sit to stands in 30 seconds)
Change in muscular strength - sit-to-stand test | The first measurement will be performed in winter 2020, with a repeat measurement approximately 3 months later in spring 2020.
  sit-to-stand test (number of sit to stands in 30 seconds)
Muscular strength - grip-strength test | One measurement at baseline
  grip-strength test (kg)
Change in muscular strength - grip-strength test | The first measurement will be performed in winter 2020, with a repeat measurement approximately 3 months later in spring 2020.
  grip-strength test (kg)
International Physical Activity Questionnaire (IPAQ) short form | One measurement at baseline
  Physical activity questionnaire to determine physical activity levels
Sun exposure questionnaire | One measurement at baseline
  Measures amount of time spent in the sun (often, occasionally, never) and what parts of the body are exposed (head, hands, arms, legs, torso) over summer, spring, autumn and winter. Also questions any summer holidays abroad, in what month, what country was visited, number of hours of sun per day and what body parts were exposed (head, hands, arms, legs, torso)
Lifestyle questionnaire | One measurement at baseline
  Measures:
  - Skin type (Fitzpatrick scale)
  Questions:
  * Questions what race they identify with
  * Holidays abroad
  * Education
  * Origin
  * Health
  * Pregnancy
  * Sun behaviours (what body parts are usually exposed to the sun, clothing, sun bathing, sunscreen use, sun bed use)
  * Smoking
  * Drinking
  * Recreational drug use
  * Knowledge around vitamin D
  * supplement use
  * Milk, egg, oily fish and liver consumption

CONTACTS AND LOCATIONS:
Locations (1):
- University of Surrey, Guildford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data from participants will be shared with researchers from partner universities (University of Surrey, University of Wollongong, University of Sao Paul and North Carolina State University)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Project data will be held for at least 6 years and all research data for at least 10 years in accordance with University policy and in accordance with the {UK} Data Protection Act (2018)
Access Criteria: Anoymised data only. Data will be shared virtually with those in the research teams at partner universities.

REFERENCES:
- [Background] Natcen.ac.uk. (2018). NatCen Social Research. [online] Available at: http://www.natcen.ac.uk/news-media/press-releases/2018/january/natcen-and-mrc-epidemiology-unit-cambridge-to-deliver-national-diet-and-nutrition-survey/ [Accessed 16 July. 2019].
- [Background] Sturges, M. & Cannell, JJ (2018). Meta-analysis questions relationship between vitamin D and bone health among the elderly. [online] The Vitamin D Council Blog & Newsletter, January 23, 2018 [Accessed 16 July. 2019].
- [Background] Wall, BF, Haylock, R, Jansen, JTM, Hillier, MC, Hart, D, Shrimpton PC (2011). Radiation Risks from Medical X-ray Examinations as a Function of the Age and Sex of the Patient. [online] https://pdfs.semanticscholar.org/d90f/22c2c119c618c6822eb094087464e5ca3c4b.pdf [Accessed 7 October 2019)
- [Background] Wilson LR, Tripkovic L, Hart KH, Lanham-New SA. Vitamin D deficiency as a public health issue: using vitamin D2 or vitamin D3 in future fortification strategies. Proc Nutr Soc. 2017 Aug;76(3):392-399. doi: 10.1017/S0029665117000349. Epub 2017 Mar 28. PMID 28347378
- [Background] Libon F, Cavalier E, Nikkels AF. Skin color is relevant to vitamin D synthesis. Dermatology. 2013;227(3):250-4. doi: 10.1159/000354750. Epub 2013 Oct 17. PMID 24134867